CLINICAL TRIAL: NCT06091644
Title: Comparison of AirAngel® vs Storz® Videolaryngoscope and Macintosh® Laryngoscope for Endotracheal Intubation Training: Prospective Randomized Crossover Study
Brief Title: The Performance of AirAngel® Videolaryngoscope
Acronym: 3D-printed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ATADEK, 2020-25/22
Record Dates: First submitted 2023-10-10; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Educational Problems; Financial Hardship
Keywords: Videolaryngoscope; 3-D printing; 3-Dimensional Printing
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of device performances in normal and difficult airway management (Other): Each endotracheal intubation (ETI) attempt could enhance the participant's experience in the next attempt. Hence, the order of use of ETI devices was randomized to avoid experience-based bias. Six subgroups were needed to determine the order in which the SMSS would use the devices based on a permutation of three because three ETI devices were planned to be used in total. Accordingly, participants were randomized into six groups using the Random Team Generator.
  Six experiment stations were set up. Normal airway manikins (NAMs) were used in the first three stations, and difficult airway manikins (DAMs) were used in the subsequent three. The interventions were to be conducted by the participants using NAMs first, followed by DAMs in the predetermined randomization order. Participants were assisted by an experienced assistant researcher in ETI during their attempts to extend the ETT, who also check the intubation accuracy with a bag valve mask (BVM) at the end of the intervention.
  Interventions: Device: AirAngel® 3D printed videolaryngoscope

INTERVENTIONS:
Device: AirAngel® 3D printed videolaryngoscope — This is a mannequin study that aims to compare a videolaryngoscope produced with 3D printing with a Storz videolaryngoscope and a Macintosh direct laryngoscope in the hands of inexperienced users in terms of ease of use, glottic imaging and intubation success.
  Other Names: Storz® videolaryngoscope and; Macintosh® laryngoscope

SUMMARY:
Video laryngoscopy (VL) have certain advantages over other techniques, such as better glottic imaging, higher intubation success in individuals with difficult airways, less force required for intubation, less cervical spine movement, and better image capturing overall. Some experts have recently suggested that the VL should be accepted and used as the standard technique for imaging in all emergency intubations, not just difficult intubations. However, VL is often not accessible in low-income countries because of its high costs. Additionally, hospitals may not be able to reach the devices even if they can cover the cost in cases where the demand is excessive.

Three dimensional (3D) printing is the technology of producing objects in 3D from an existing or designed digital file. This rapidly developing technology is already used in many areas of daily life and has also been widely used in medical applications. 3D printers produce many expensive medical materials and devices at lower costs, enable personalized modeling (implants and prostheses), tissue cultures, and surgical planning, and can also be used as educational material. One of these applications is 3D-printed VL (3D-PVL), which has become prominent in pandemic conditions. A 3D-PVL can be obtained for only 6-30 United States dollars (USD) compared to a VL that costs thousands of US dollars.

Moreover, a study comparing 3D-PVL with standard VL in difficult airway management for experienced practitioners demonstrated comparable success rates in both devices. Furthermore, the VL created by modifying a Macintosh® laryngoscope (MCL) with an endoscope camera was reported superior to the standard MCL and comparable to the standard VL in the hands of experienced users. However, the literature presented no study that evaluated the efficiency of 3D-PVLs in inexperienced practitioners. Herein, our study aimed to investigate the effectiveness of 3D-PVLs in acquiring endotracheal intubation (ETI) skills in senior medical school students who are inexperienced users and compare 3D-PVL with standard MCL and VL.

DETAILED DESCRIPTION:
Materials The globally accessible AirAngel® 5.5-mm standard adult laryngoscope model was chosen as the 3D-PVL blade model. AirAngel® is a 3D-PVL model produced with 3D printing technology, the digital file of which has been opened to public access by its designers, which has a hyper-angulated blade and allows transferring the images to devices such as a phone, computer, or tablet with an integrated endoscope camera. The AirAngel® 3D 5.5-mm standard adult laryngoscope model was printed with 3D printer at Acibadem Mehmet Ali Aydinlar University Incubation Center in 80% density and as five layers from polylactic acid (PLA) material. The indentation at the end of the printed laryngoscope was suitable for integrating a 5.5-mm diameter camera (endoscope). The PLA material used in printing costs approximately 6 USD.

We mounted a 5.5-mm diameter, light-emitting diode (LED)-illuminated, International Protection Code (IP)67-certified, and water-resistant endoscope camera with a resolution of 640 × 480 pixels equipped with a 1/9 inch complementary metal oxide semiconductor sensor and 1-m long universal serial bus (USB) connection to the printed laryngoscope for approximately 9 USD. The created 3D-PVL was connected to a smart phone compatible with USB On-The-Go, which is a feature that allows the phone to be used as a host allowing the use of other USB devices, with a 6.67-inch in-plane switching liquid crystal display with a resolution of 1080 × 2400 full high definition+ pixels. A smart phone-supported 3D-PVL was obtained in this way.

A standard MCL and Storz® VL (SVL) monitor was selected as the DL and VL devices to be compared with 3D-PVL, respectively. A size 3 Macintosh blade, which is the most commonly used in adults and compatible with 3D-PVL dimensions and design, was preferred for both MCL and SVL.

The tongue of the manikin was fully inflated with 10 mL of air when the manikin was being used as a difficult airway manikin (DAM), and the cervical spine screw was fully tightened to reduce head extension. No modifications were made when the manikin was used as a normal airway manikin (NAM). An endotracheal tube (ETT) with a standard 7.5-mm inner diameter was chosen. The stylet was placed in the ETT before the intervention. A new ETT and stylet were used in each intervention. Additionally, the ETTs were lubricated before each intervention.

Participants The study participant consisted of senior students enrolled in Acibadem Mehmet Ali Aydinlar University Faculty of Medicine. The study was conducted at the Center of Advanced Simulation and Education (CASE) laboratory. The senior medical school students (SMSS) were invited via e-mail by the medical education coordination office of the university from November 2020 to January 2022. SMSS were invited four times in total, twice in each academic year. Informed consent and study plan were shared within the invitation e-mail. The e-mail stated that this study would not be graded, it would not have any effect on school success, participation is not compulsory, and they can participate in the study by making an appointment with CASE at any time during the academic year.

The sample size was calculated using the G*Power Software® version 3.1.9.2 as follows based on the statistical comparison conducted according to the referenced publication. Type-1 error and power of the test were chosen as 5% and 95%, respectively. Consequently, the targeted sample size was calculated as 126 considering randomization. The applications received after a sufficient number of students applied to the study were rejected, and no more students were recruited.

SMSS routinely participate in the standardized airway training module during sixth-grade medical school education. ETI training is given with both standard MCL and VL in this module. Thus, users who received standardized training were the SMSS included in the study. Additionally, participants were asked about any experience in intubating a patient and none had any experience. A 30-min training video was prepared that indicated the differences between DL and VL, introduced DAMs and NAMs, and demonstrated ETI practices. All participants were required to watch this training video before the intervention.

Randomization Each ETI attempt could enhance the participant's experience in the next attempt. Hence, the order of use of ETI devices was randomized to avoid experience-based bias. Six subgroups were needed to determine the order in which the SMSS would use the devices based on a permutation of three because three ETI devices were planned to be used in total. Accordingly, participants were randomized into six groups using the Random Team Generator. Each group included 21 participants.

Study Protocol Six experiment stations were set up. Each table was ensured to have one airway manikin. NAMs were used in the first three stations, and DAMs were used in the subsequent three. The interventions were to be conducted by the participants using NAMs first, followed by DAMs in the predetermined randomization order. Participants were assisted by an experienced assistant researcher in ETI during their attempts to extend the ETT, who also check the intubation accuracy with a bag valve mask (BVM) at the end of the intervention.

Each participant was given 3 min before each intervention to be prepared for the device and manikin. It was aimed that the participants would not feel pressed for time and would not attempt to intubate quickly. To this end, 1 min was given to complete the intubation attempt. The intervention was started as the participant said, "I am ready," and the assistant researcher vented the ETT with the BVM as the participant said, "I am done," after he/she was sure that he/she had placed the ETT. The intubation time was assessed as the time elapsed between placing the laryngoscope in the mouth and the ventilation of the lungs or stomach. The intubation attempt was terminated although it was not completed yet and considered unsuccessful when the intubation time was over 1 min. Accurate ETT placement was evaluated by visual confirmation of the swelling of the lungs on the manikin. The intubation attempt was considered unsuccessful if the manikin's stomach was filled with air. Conversely, the intubation attempt was considered successful if one or both lungs were filled with air.

An unsuccessful intubation attempt is considered a failure of three or more intubation attempts by an experienced user, or the failure of the patient to maintain an airway when a permanent airway is required immediately. Conservative airway management maneuvers should be limited to 2-3 min because irreversible cerebral anoxia occurs within minutes. The maximum recommended duration of an intubation attempt is 30 s although with no precise definition of an unsuccessful intubation attempt in the literature. Intubation should continue after the patient is ventilated with BVM if the intubation period exceeds 30 s. Hence, intubation attempts that lasted longer than 30 s were considered unsuccessful, although the participants were given 1 min to complete the intubation. Thus, only the intubation attempts that lasted ≤30 s, in which the ETT was accurately placed in the trachea, and the lungs were ventilated were considered successful. The rate of successful intubation attempts was calculated based on the intubation attempts deemed successful according to the said criteria.

The participants were asked to evaluate the ease of use of the device with a 5-point (from very easy to very difficult) Likert-type scale and to what extent they could view the vocal cords during the intervention according to the Cormack-Lehane classification, which was provided to the SMSS with visual material in the form a Likert-type scale, after each intubation attempt. Thus, intubation times, ease of use scores, Cormack-Lehane grades, rates of accurate placement of ETT, and rates of successful intubation attempts were measured at the end of each intubation attempt with DAM or NAM using any of the three laryngoscopy devices.

ELIGIBILITY:
Inclusion Criteria:

Being senior medical students Not having received endotracheal intubation training

Exclusion Criteria:

Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Effectiveness of 3D printed videolaryngoscope | Two years
  It is a mannequin study that aims to compare a videolaryngoscope produced with 3D printing with a Storz videolaryngoscope and a Macintosh direct laryngoscope in the hands of inexperienced users in terms of intubation success. Accurate ETT placement was evaluated by visual confirmation of the swelling of the lungs on the manikin. The intubation attempt was considered unsuccessful if the manikin's stomach was filled with air. Conversely, the intubation attempt was considered successful if one or both lungs were filled with air. An unsuccessful intubation attempt is considered a failure of three or more intubation attempts by an experienced user, or the failure of the patient to maintain an airway when a permanent airway is required immediately.

SECONDARY OUTCOMES:
The effectiveness of using a 3D printed videolaryngoscope during endotracheal intubation training. | Two years
  Access to VLs is restricted due to their high cost, and we investigated whether a 3D printed videolaryngoscope could be used instead of these devices in intubation training. The participants were asked to evaluate the ease of use of the device with a 5-point (from very easy to very difficult) Likert-type scale and to what extent they could view the vocal cords during the intervention according to the Cormack-Lehane classification, which was provided to the SMSS with visual material in the form a Likert-type scale, after each intubation attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Kayayurt, Ass Prof, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pieters BMA, Maas EHA, Knape JTA, van Zundert AAJ. Videolaryngoscopy vs. direct laryngoscopy use by experienced anaesthetists in patients with known difficult airways: a systematic review and meta-analysis. Anaesthesia. 2017 Dec;72(12):1532-1541. doi: 10.1111/anae.14057. Epub 2017 Sep 22. PMID 28940354
- [Background] Maruyama K, Yamada T, Kawakami R, Hara K. Randomized cross-over comparison of cervical-spine motion with the AirWay Scope or Macintosh laryngoscope with in-line stabilization: a video-fluoroscopic study. Br J Anaesth. 2008 Oct;101(4):563-7. doi: 10.1093/bja/aen207. Epub 2008 Jul 25. PMID 18660500
- [Background] Zaouter C, Calderon J, Hemmerling TM. Videolaryngoscopy as a new standard of care. Br J Anaesth. 2015 Feb;114(2):181-3. doi: 10.1093/bja/aeu266. Epub 2014 Aug 23. No abstract available. PMID 25150988
- [Background] Lambert CT, John SC, John AV. Development and performance testing of the low-cost, 3D-printed, smartphone-compatible 'Tansen Videolaryngoscope' vs. Pentax-AWS videolaryngoscope vs. direct Macintosh laryngoscope: A manikin study. Eur J Anaesthesiol. 2020 Nov;37(11):992-998. doi: 10.1097/EJA.0000000000001264. PMID 32675700
- [Background] Cook TM, Kelly FE. A national survey of videolaryngoscopy in the United Kingdom. Br J Anaesth. 2017 Apr 1;118(4):593-600. doi: 10.1093/bja/aex052. PMID 28403414
- [Background] Coles-Black J, Chao I, Chuen J. Three-dimensional printing in medicine. Med J Aust. 2017 Aug 7;207(3):102-103. doi: 10.5694/mja16.01073. No abstract available. PMID 28764624